CLINICAL TRIAL: NCT03932721
Title: EXpanded Combination of Evolocumab Plus Empagliflozin on Diabetes: EXCEED-BHS3 Trial
Acronym: EXCEED-BHS3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Coordinator of the Brazilian Heart Study Group, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Exceed
Record Dates: First submitted 2019-04-12; First posted 2019-05-01 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Dyslipidemia Associated With Type II Diabetes Mellitus; Diabetes Mellitus, Type 2; Hypertension Arterial
Keywords: Dyslipidemia; Diabetes Mellitus, Type 2; Hypertension Arterial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to evolocumab (140 mg every two weeks) on top of the standard of care, SOC therapy ( SGLT2 inhibitors, maximal statin dose and ideal control of blood glucose (HbA1c 6.5% to 7%) and blood pressure (SBP <140 mm Hg). Or to the exclusive use of the SOC therapy.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evolocumabe (Active Comparator): Patients with T2DM treated with the standard of care (SGLT2 inhibitors, maximal statin dose and ideal control of blood glucose and blood pressure) AND evolocumab (anti-PCsk9).
  Interventions: Drug: Evolocumab 140 MG/ML
- Control (No Intervention): Patients with T2DM treated exclusive with the standard of care (SGLT2 inhibitors, maximal statin dose and ideal control of blood glucose and blood pressure).

INTERVENTIONS:
Drug: Evolocumab 140 MG/ML — Evolocumab is a fully human monoclonal antibody that inhibits proprotein convertase subtilisin/kexin type 9 (PCSK9). PCSK9 is a protein that targets LDL receptors for degradation and thereby reduces the liver's ability to remove LDL-C.
  Other Names: Control
  Arms: Evolocumabe

SUMMARY:
Based on the current evidence, empagliflozin could reduce cardiovascular morbidity and mortality in Diabetes Mellitus Type 2 (T2DM). Anti-PCSK9 therapy (evolocumab) can reduce the major cardiovascular events incidence in secondary prevention individuals, some of them presenting T2DM. The beneficial effect of the combined use of these two agents in T2DM remains unknown. Evaluating the effect of evolocumab on top of the best of care therapy for T2DM, including empaglifozin, on endothelial function may indicate the existence of some benefit related to cardiovascular outcomes.

DETAILED DESCRIPTION:
Study design: Randomized, parallel-group, open, comparative, prospective clinical study.

Eligibility criteria will be: T2DM between 40 and 70 years old; adequate glycemic control; (HbA1c 7 to 9%) after run-in phase; adequate blood pressure control (SBP ≤ 140 mm Hg); maximal tolerated dose of statins and LDL-C between 70 and 100 mg/dL.

Volunteers' convocation -Investigators will announce in radio, television and newspapers inviting volunteers with T2DM for this study. Those who contact us with an interest in participating by email or whatsapp will be enrolled for the first telephone screening evaluation. These volunteers will be contacted by phone and after a detailed explanation about the objectives, procedures, and shared responsibilities between the parties those willing to participate will be summoned to a Screening Visit (SV) in which inclusion and exclusion criteria will be further verified. The screening FMD will be measured in this occasion.

Run-In - In the following two weeks after the screening visit, patients must return to another consultation in which antidiabetic, antihypertensive and lipid-lowering therapies adjustment will be performed. The adjustment period must be ended at 16 weeks and if this is not so patients will be excluded.

Pre-randomization exams - In the two weeks preceding the Randomization Visit, patients will undergo laboratory tests (urea, creatinine, blood glucose, total cholesterol, HDL-c, LDL-col, HbA1c, triglycerides).

Randomization Phase - At the Randomization Visit (RV): Blood samples will be collected and frozen at -250oC for laboratory analysis at the end of the trial. Patients will be submitted to a protocol for assessing endothelial function (FMD).

Thereafter, patients will be assigned to evolocumab (140 mg every two weeks) on top of the standard of care therapy (SOC) or to the exclusive use of the SOC.

At thirty days (Visit 1), 4 weeks (Visit 2), 8 weeks (Visit 3), 12 weeks (Visit 4) and 16 weeks (Visit 5) post-randomization, patients will be seen at the outpatient clinic for evaluation of overall clinical status, treatment adherence through count of tablets, adverse events and use of concomitant medications. Evolocumab will be administered at study center every 15 days.

At the Visits 3 and 5, FMD will be reassessed and new blood samples will be collected and stored.

Protocol of Endothelial Function Assessment: Brachial artery measurements will be performed using a high-resolution ultrasound (Vivid q, GE Medical System, Milwaukee, WI, USA), obtained by physicians with long experience in this exam. The procedure will take place after over-night fasting and withdrawal of any vasoactive medications for the previous 24 hours. After ten minutes of quiet resting in a room with controlled temperature (around 25°C), the brachial artery will be located above the antecubital fossa, and a longitudinal image of 6 to 8 cm of the artery will be considered as the baseline scan. A size appropriate blood pressure cuff will be placed around the forearm and inflated up to 50 mmHg above the systolic blood pressure for five minutes and the cuff will be then deflated. The FMD scan will be obtained for 5 minutes. An adjustable stereotaxic clamp will stabilize the probe. Percentage change in diameter for FMD will be calculated in relation to the respective baseline scans. Video clips will be recorded for 1 minute before cuff inflation and then restarted 1 minute before cuff deflation until 5 minutes after deflation.

Laboratory methods - At randomization, 8th and 16th week, blood samples will be obtained for measuring: Glucose, C Reactive protein, HbA1c, triglycerides. At the same time points, blood samples will also be obtained before and after the two FMD measurements (pre and post-ischemia) and will be assessed for VCAM-1 and NO. NO and its metabolites, i.e. nitrite and nitrate (NOx), will be measured by an NO chemiluminescence analyzer (model NOA, Sievers Instruments, Boulder, CO). Isoprostane will be measured by ELISA at randomization, 8th and 16th week of therapy.

Lipoproteins fractions isolation by gradient ultracentrifugation - Lipid profile will be assessed at admission, at the 8th week and at the 16th week by gradient ultracentrifugation. VLDL, LDL (1 to 5 subfractions) and HDL (2b to 3a subfractions) will be isolated through density gradient ultracentrifugation using a SW41Ti rotor. Isolated lipoproteins content in cholesterol will be measured using commercially available enzymatic kits total cholesterol (TC) (CHOD-PAP, Roche Diagnostics® reagents, Mannheim, Germany)], in the microplate reader Power Wave XS (BioTek®, Winooski, USA).

Sample size and Statistical Analysis - Investigators are not aware of any studies that have evaluated the effect of evolocumab or other anti-PCSK9 antibody on FMD. However, two trials with similar characteristics to this design were performed testing the effects of atorvastatin 80 mg/day or rosuvastatin 40 mg/day on conventional FMD. A difference of 3% after treatment was noticed in both trials, with a mean pre-treatment value of 5.5% and a standard deviation of 3.9%.

Considering an alpha value of 0.05 and beta of 90%, this study would require 49 patients per arm. Accounting for dropout and exclusion of patients during the pre-randomization phase and the trial, investigators propose 12% of drop-off, equivalent to 110 patients, 55 in each arm. Investigators used G-Power to calculate sample size. Covariance analysis (ANCOVA) will be used to evaluate the effect of treatments on the mean change in FMD at the 16th week, the primary endpoint. The assumptions of ANCOVA models (linearity, distribution normality and equal variance) will be verified using histograms, normal probability plots and residual scatter plots. Age, gender and baseline FMD values will be included as covariables in all ANCOVA models. The adjustment for the baseline values is intended to adjust for the possible regression to the mean bias. Non-normal continuous variables will be transformed by logarithm to correct dispersion. If after transformation they persist not normal, these variables will be analyzed by the Kruskal-Wallis test.

Statistical significance in the secondary endpoints will only be considered if the primary outcome is statistically significant. All of the exploratory endpoints will be reported with 95% CIs. In order to assure the quality of measurements, inter- and intra-patient variability of FMD will be obtained in a set of patients from the screening phase of the study.

Randomization - Stratified randomization will be used in this study. Individuals will be allocated in one of the four groups generated by the following parameters that could interfere on endothelial function: gender and age (40 -55 or 56 - 70 years old).

Adverse Events will be collected from time of signature of informed consent, throughout the treatment period until the last visit. Serious Adverse Events (SAEs) will be recorded from the time of informed consent.

Reporting of serious adverse events - All SAEs have to be reported in the CRF, whether or not considered causally related to the investigational product or to the study procedure(s). According to local sanitary (ANVISA) and ethics (CEP/CONEP) regulations, SAEs must be reported to the regulatory authority and AMGEN at the same time.

ELIGIBILITY:
Inclusion Criteria:

* T2DM between 40 and 70 years old;
* Adequate glycemic control (HbA1c 7 to 9%) after run-in phase;
* Adequate blood pressure control (SBP ≤ 140 mm Hg)
* Maximal tolerated dose of statins and LDL-C between 70 and 100 mg/dL.

Exclusion Criteria:

* HbA1c > 9% after run-in phase;
* Hospitalization for unstable angina or acute myocardial infarction within 6 months prior to enrolment;
* Acute stroke or transient ischemic attack (TIA) within 6 months prior to enrolment;
* Less than two months post coronary artery revascularization;
* BP ≥ 140 x 90 after anti-hypertensive medication adjustment;
* FMD <2% or > 10% at the time of randomization;
* Triglycerides > 500 mg/dL;
* Known allergy to any of the study drugs;
* Severe coronary artery disease or heart failure;
* Systemic inflammation (C-reactive protein ≥ 5 mg/dL);
* Pregnancy or women during reproductive age;
* Active smoking or stopped smoking less than six months ago;
* Participation in other clinical studies or whose participation ended less than six months -ago.
* Use of SGLT2i or GLP-1a in the last sex months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Difference in the percentage change in flow mediated dilation (FMD) | 16 weeks
  Difference in the change in flow mediated dilation (FMD) between the randomization visit and at 16 weeks of treatment. Brachial artery measurements will be performed using a high-resolution ultrasound obtained by physicians with long experience in this exam. The FMD scan will be measured on Video clips recorded from 1 minute before cuff inflation to 5 minutes after deflation. Percentage change in diameter for FMD will be calculated in relation to the respective baseline scans.

SECONDARY OUTCOMES:
Difference in the percentage change in FMD reserve | 16 weeks
  Difference in the change in FMD reserve (change after ischemia/reperfusion) between the randomization visit and at 16 weeks of treatment. FMD reserve will be estimated by the difference between rest and post-ischemia assessment. Briefly, FMD will be assessed at rest and repeated after 30 minutes of brachial ischemia followed by 15 minutes of reperfusion. The percentage difference between baseline and post-ischemia FMD will be considered as FDM reserve.

OTHER OUTCOMES:
Difference in the change of plasma NO in mmol/L | 16 weeks
  Difference in the change of plasma NO in mmol/L after FMD at the randomization visit and at 16 weeks of treatment.
Difference in the change of plasma VCAM-1 in pg/mL | 16 weeks
  Difference in the change of plasma VCAM-1 in pg/mL at the randomization visit and at 16 weeks of treatment.
Difference in the percentage change in FMD from randomization to 8 weeks of treatment. | 8 weeks
  Difference in the percentage change in FMD between the randomization visit and at 8 weeks of treatment.
Difference in the percentage change in FMD reserve from randomization to 8 weeks of treatment. | 8 weeks
  Difference in the change in FMD reserve between the randomization visit and at 8 weeks of treatment.
Difference in the change in plasma isoprostane in pg/mL from randomization to 16 weeks of treatment. | 16 weeks
  Difference in the change in plasma isoprostane in pg/mL between the randomization visit and at 16 weeks of treatment.
Difference in the percentage change of LDL subfractions from randomization to 16 weeks of treatment. | 16 weeks
  Difference in the percentage change of the distribution of LDL subespecies between the randomization visit and at 16 weeks of treatment.
Difference in the Change of Ambulatorial Blood Pressure (mm Hg) from randomization to 16 weeks of treatment. | 16 weeks
  Difference in the Change of Ambulatorial Blood Pressure (mm Hg) between the randomization visit and at 16 weeks of treatment.
Difference in Plasma C-Reactive Protein Change in mg/dL from randomization to 16 weeks of treatment. | 16 weeks
  Difference in Plasma C-Reactive Protein Change in mg/dL between treatments from randomization visit to 16 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, MD,Phd, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Centro de Pesquisa Clinica - FCM/Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breder I, Cunha Breder J, Bonilha I, Munhoz DB, Medorima STK, Oliveira DC, do Carmo HR, Moreira C, Kontush A, Zimetti F, Zanotti I, Carvalho LSF, Nadruz W, Muscelli E, Quinaglia T, Sposito AC; EXCEED-BHS3 Trial Investigator. Rationale and design of the expanded combination of evolocumab plus empagliflozin in diabetes: EXCEED-BHS3 trial. Ther Adv Chronic Dis. 2020 Sep 28;11:2040622320959248. doi: 10.1177/2040622320959248. eCollection 2020. PMID 33062236